CLINICAL TRIAL: NCT05655013
Title: Treatment With Zoledronate Subsequent to Denosumab in Osteoporosis 2 (ZOLARMAB2)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anne Sophie Sølling, MD, PhD, Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01.12.2022
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Part 1: 1-year randomized open label, interventional study in 200 postmenopausal women.
  Part 2: 2-year randomised, double-blind, interventional study in the women completing part 1.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First part (year 1): groups 1+2 (Active Comparator): Zoledronate will be administered as an infusion six months after the last injection of denosumab followed by zoledronate infusions 3 and 6 months thereafter
  Interventions: Drug: Zoledronate
- First part (year 1): groups 3+4 (Active Comparator): Zoledronate will be administered as an infusion six months after the last injection of denosumab followed by zoledronate infusions when bone turnover is increased (s-carboxy-terminal collagen crosslinks (p-CTX) > 0.4 ug/l which corresponds to the upper 50 % of the normal range for premenopausal women).
  Interventions: Drug: Zoledronate
- Second part (year 2-3): groups 1+3 (Active Comparator): Patients will receive yearly infusions of zoledronate 5 mg
  Interventions: Drug: Zoledronate
- Second part (year 2-3): groups 2+4 (Placebo Comparator): Patients will receive yearly infusions of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronate — zoledronate 5 mg
  Arms: First part (year 1): groups 1+2; First part (year 1): groups 3+4; Second part (year 2-3): groups 1+3
Drug: Placebo — isotonic saline 100 mL
  Arms: Second part (year 2-3): groups 2+4

SUMMARY:
The aims of ZOLARMAB2 are fourfold. First, the investigators want to investigate if multiple infusions of zoledronate can prevent the rebound activation of bone turnover and the subsequent bone loss in patients previously treated with denosumab and if there is difference between infusing zoledronate at fixed time-points after the last injection of denosumab or when bone turnover is increased.

Second, the investigators want to investigate if bone loss will resume after controlling the rebound activation of bone turnover during the first year after denosumab discontinuation and if this can be prevented by yearly infusions of zoledronate.

Third, the investigators want to investigate the underlying pathophysiological mechanisms by investigating biochemical markers, osteoclast and osteoblast activation signals in the bone and bone marrow, and the pool of preosteoclasts/mature osteoclasts before and after treatment with zoledronate.

Fourth, the investigators want to investigate the effect of denosumab discontinuation on muscle mass and muscle strength and on insulin sensitivity.

DETAILED DESCRIPTION:
This study has two parts. The first part (year 1) is a randomized open label, interventional study in 200 postmenopausal women investigating if treatment with zoledronate prevents bone loss after denosumab treatment. Zoledronate will be administered as an infusion six months after the last injection of denosumab followed by zoledronate infusions 3 and 6 months thereafter (groups 3+4) or followed by zoledronate infusions when bone turnover is increased (p-carboxy-terminal collagen crosslinks (p-CTX) > 0.4 ug/l which corresponds to the upper 50 % of the normal range for premenopausal women) (groups 1+2). Fifty patients will be randomised to each group. The patients in groups 1+2 will be monitored and if (p-CTX) is above 0.4 ug/l at month 3 or 6 zoledronate will be administered. If a patient in groups 3+4 experiences an osteoporotic clinical vertebral or hip fracture, zoledronate will be administered irrespective of p-CTX.

The second part is a 2-year randomised, double-blind, interventional study in the women completing part 1. Patients in groups 1+3 will receive yearly infusions of zoledronate 5 mg and patients in groups 2+4 will receive yearly infusions of placebo.

The patients will be monitored with DXA of the hip and spine 3, 6, 12, 24, and 36 months after baseline. Zoledronate will be administered to the patients allocated to the placebo group during phase 2 if BMD decreases more than 5% at the lumbar spine, total hip or femoral neck after months 12.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal for at least two years)
* Age ≥ 40 years
* Treatment for at least two years with denosumab
* Last denosumab injection less than six months ago
* At least 2 lumbar vertebrae that can be evaluated by DXA

Exclusion Criteria:

* Low-energy vertebral fracture within the last ten years
* Multiple low-energy vertebral fractures (> 3) at any time
* Low-energy hip fracture within the last 12 months
* BMD T-score < -2.5 (lumbar spine, total hip or femoral neck)
* Zoledronate treatment for more than three years prior to denosumab treatment within the last ten years
* Alendronate treatment for more than three years prior to denosumab treatment within the last five years or for more than five years within the last 10 the years
* Treatment with other bisphosphonates (risedronate, ibandronate) for more than three years prior to denosumab treatment within the last five years
* Diabetes Mellitus
* Ongoing treatment with systemic glucocorticoids
* Metabolic bone disease (for example osteogenesis imperfecta, Paget's disease of bone)
* Hormone replacement therapy
* Active cancer within the last 5 years with the exception of basal cell skin cancer
* Estimated glomerular filtration rate (eGFR) ≤ 35 mL/min
* Contraindications for zoledronate according to the SPC
* Unable to read and understand Danish
* Immobility

Ages: 40 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in lumbar spine bone mineral density (BMD) | After 12 and 36 months.
  Change in lumbar spine BMD after 12 and 36 months.
The proportion of patients who fails to maintain bone mineral density (BMD) | After 12 months.
  The proportion of patients (%) with significant decrease in BMD (≥ 3 % BMD loss at the lumbar spine or ≥ 5 % BMD loss at the femoral neck or total hip) after 12 months.

SECONDARY OUTCOMES:
Changes in total hip and femoral neck bone mineral density (BMD) | After 12 and 36 months.
  Changes in total hip and femoral neck BMD after 12 and 36 months.
Changes in trabecular bone volume fraction (bone volume/tissue volume, BV/TV) and cortical porosity measured by high-resolution peripheral quantitative computed tomography (HR-pQCT) | After 12 and 36 months.
  Mean percent change in trabecular bone volume fraction and cortical porosity measured by HR-pQCT at the radius and tibia after 12 and 36 months.
Changes in carboxy-terminal collagen crosslinks (CTX) and procollagen type I N-terminal propeptide (PINP) | After 3, 6, 12, 24 and 36 months.
  Changes in CTX and PINP after 3, 6, 12, 24 and 36 months.
Morphometric vertebral fractures | After 12 and 36 months.
  Morphometric vertebral fractures assessed by vertebral fracture assessment (VFA) after 12 and 36 months or by spinal x-ray if clinical suspicion of vertebral fracture.
Serum RANKL/OPG, tartrate-resistant acid phosphatase type 5b (TRAcP-5b), sclerostin and Dickkopf-1 (Dkk-1) | Baseline and after 1, 3, 6 and 12 months
  Serum RANKL/OPG, tartrate-resistant acid phosphatase type 5b (TRAcP-5b), sclerostin and Dickkopf-1 (Dkk-1) at 0, 1, 3, 6 and 12 months
Molecular bone histology | Baseline and after 3 months
  Molecular bone histology of accumulating osteoclast activation sites and pre-osteoclasts as well as single-nucleus transcriptomics on jamshidi biopsies at baseline in a total of 100 patients from groups 1 and 2 and in up to 15 participants in groups 1 and 2 at month 3 with a strong rebound response (p-CTX > 0.6 ug/l).
Osteoclasts | Baseline
  Osteoclasts differentiation, fusion, function, and response to zoledronate in cultures derived from peripheral blood at baseline from groups 1 and 2. 30 patients will be recruited from each group, hence 60 patients.
Epigenetic marker analysis | Baseline
  Epigenetic marker analysis with special focus on genes involved in osteoclast activation, differentiation, fusion, function and response to ZOL. Samples collected at baseline from all participants.
Muscle mass and muscle strength | Baseline and after 3 and 12 months
  Muscle mass assessed by whole-body DXA and muscle strength assessed by handgrip strength and muscle strength over the knee and elbow joints. A total of 100 patients from groups 1 and 2 will be investigated at baseline month 3 and 12.
Insulin sensitivity | Baseline and after 3, 12, 18, 24 and 36 months
  Insulin sensitivity assessed by Hb1Ac, HOMA-IR, OGTT and advanced glycation end products (AGEs).

CONTACTS AND LOCATIONS:
Overall Officials: Bente Langdahl, MD, Professor, DMSc, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No